CLINICAL TRIAL: NCT00488436
Title: SMD/ATG-CSA: Antithymocyte Globulin and Cyclosporine in Treating Low Risk Patients With Myelodysplastic Syndrome
Brief Title: Antithymocyte Globulin and Cyclosporine in Treating Low Risk Patients With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Pethema, pethema
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMD/ATG-CSA/2002
Record Dates: First submitted 2007-06-19; First posted 2007-06-20 (Estimated); Last update posted 2008-11-19 (Estimated); Status verified 2008-11

CONDITIONS: Myelodysplastic Syndrome
Keywords: Myelodysplastic Syndrome; Antithymocyte Globulin; Cyclosporine
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Antilymphocyte Serum; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Antithymocyte globulin
Drug: Cyclosporine

SUMMARY:
The different mechanisms of action between Antithymocyte globulin and cyclosporine can improve the effectivity when both are used in combination in patients with myelodysplastic syndrome.

DETAILED DESCRIPTION:
Patients are treated with:

Antithymocyte globulin (Timoglobulin SangStat)

* 2,5 mg/kg/day IV over 8 hours on days 1-4
* Total dose: 10 mg/kg
* Calculated dose adjusted to ideal weight
* Especial considerations:

Paracetamol 1 gr (oral or IV) Dexclorfeniramine 5 mg IV Methylprednisolone 1 mg/kg IV 30 minutes before Timoglobulin and repeat if necessary at 4 hours - Platelet transfusion if platelet count is < 50 x 109/L

Cyclosporine (Sandimmun Neoral)

-2,5 mg/kg/12 h over 3 months

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of low or intermediate risk myelodysplastic syndrome (MDS) (or high risk patient not eligible to intensive chemotherapy or for bone marrow transplantation), excluding chronic myelomonocytic leukemia
* At less one of two following conditions:
* Transfusion dependence: 1)Packed red blood cell transfusions greater than 2 times; 2)Untransfused hemoglobin level no greater than 10 g/dL; 3)Platelet transfusions greater than 1 time
* Infection grade III or IV secondary to neutropenia
* ECOG < or = 2

Exclusion Criteria:

* Chronic myelomonocytic leukemia
* Creatinine greater than 2 mg/dl
* Bilirubin greater than 2.5 mg/dl
* History of heart failure
* History of allergy to rabbit proteins

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2002-05; Primary Completion 2007-06 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Compare the efficacy and toxicity of antithymocyte globulin and cyclosporine in patients with low risk myelodysplastic syndrome | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Sanz Guillermo, Dr, Study Director — Hospital La Fe de Valencia; Julia Antonio, Dr, Study Director — Hospital Vall d'Hebron Barcelona
Locations (11):
- Spain (11):
  - Hospital de Cabueñes, Asturias
  - Hospital germans Trias i Pujol, Badalona
  - Hospital de Basurto, Bilbao
  - Hospital Ntra Sra del Rossell, Cartagena
  - Hospital Materno Infantil de Las Palmas, Las Palmas de Gran Canaria
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Morales Messeguer, Murcia
  - Hospital de Navarra, Pamplona
  - Hospital Arnau de Vilanova, Valencia
  - Hospital Dr Pesset, Valencia
  - Hospital Clinico Universitario, Zaragoza

REFERENCES:
- [Background] Sugawara T, Endo K, Shishido T, Sato A, Kameoka J, Fukuhara O, Yoshinaga K, Miura A. T cell-mediated inhibition of erythropoiesis in myelodysplastic syndromes. Am J Hematol. 1992 Dec;41(4):304-5. doi: 10.1002/ajh.2830410425. No abstract available. PMID 1288301
- [Background] Molldrem JJ, Jiang YZ, Stetler-Stevenson M, Mavroudis D, Hensel N, Barrett AJ. Haematological response of patients with myelodysplastic syndrome to antithymocyte globulin is associated with a loss of lymphocyte-mediated inhibition of CFU-GM and alterations in T-cell receptor Vbeta profiles. Br J Haematol. 1998 Sep;102(5):1314-22. doi: 10.1046/j.1365-2141.1998.00920.x. PMID 9753062
- [Background] Smith MA, Smith JG. The occurrence subtype and significance of haemopoietic inhibitory T cells (HIT cells) in myelodysplasia: an in vitro study. Leuk Res. 1991;15(7):597-601. doi: 10.1016/0145-2126(91)90028-r. PMID 1830630
- [Background] Young NS. The problem of clonality in aplastic anemia: Dr Dameshek's riddle, restated. Blood. 1992 Mar 15;79(6):1385-92. No abstract available. PMID 1547338
- [Background] Jonasova A, Neuwirtova R, Cermak J, Vozobulova V, Mocikova K, Siskova M, Hochova I. Cyclosporin A therapy in hypoplastic MDS patients and certain refractory anaemias without hypoplastic bone marrow. Br J Haematol. 1998 Feb;100(2):304-9. doi: 10.1046/j.1365-2141.1998.00551.x. PMID 9488617
- [Background] Epperson DE, Nakamura R, Saunthararajah Y, Melenhorst J, Barrett AJ. Oligoclonal T cell expansion in myelodysplastic syndrome: evidence for an autoimmune process. Leuk Res. 2001 Dec;25(12):1075-83. doi: 10.1016/s0145-2126(01)00083-2. PMID 11684279
- [Background] Maciejewski JP, Follmann D, Nakamura R, Saunthararajah Y, Rivera CE, Simonis T, Brown KE, Barrett JA, Young NS. Increased frequency of HLA-DR2 in patients with paroxysmal nocturnal hemoglobinuria and the PNH/aplastic anemia syndrome. Blood. 2001 Dec 15;98(13):3513-9. doi: 10.1182/blood.v98.13.3513. PMID 11739151
- [Background] Molldrem JJ, Caples M, Mavroudis D, Plante M, Young NS, Barrett AJ. Antithymocyte globulin for patients with myelodysplastic syndrome. Br J Haematol. 1997 Dec;99(3):699-705. doi: 10.1046/j.1365-2141.1997.4423249.x. PMID 9401087
- [Background] Greenberg P, Cox C, LeBeau MM, Fenaux P, Morel P, Sanz G, Sanz M, Vallespi T, Hamblin T, Oscier D, Ohyashiki K, Toyama K, Aul C, Mufti G, Bennett J. International scoring system for evaluating prognosis in myelodysplastic syndromes. Blood. 1997 Mar 15;89(6):2079-88. PMID 9058730
- [Background] Bennett JM, Catovsky D, Daniel MT, Flandrin G, Galton DA, Gralnick HR, Sultan C. Proposals for the classification of the myelodysplastic syndromes. Br J Haematol. 1982 Jun;51(2):189-99. PMID 6952920
- [Background] Cheson BD, Bennett JM, Kantarjian H, Pinto A, Schiffer CA, Nimer SD, Lowenberg B, Beran M, de Witte TM, Stone RM, Mittelman M, Sanz GF, Wijermans PW, Gore S, Greenberg PL; World Health Organization(WHO) international working group. Report of an international working group to standardize response criteria for myelodysplastic syndromes. Blood. 2000 Dec 1;96(12):3671-4. PMID 11090046
- [Background] Cheson BD, Bennett JM, Kantarjian H, Schiffer CA, Nimer SD, Lowenberg B, Stone RM, Mittelman M, Sanz GF, Wijermans PW, Greenberg PL. Myelodysplastic syndromes standardized response criteria: further definition. Blood. 2001 Sep 15;98(6):1985. doi: 10.1182/blood.v98.6.1985. No abstract available. PMID 11535540
- See also: Spanish association of Haematology — http://www.aehh.org